CLINICAL TRIAL: NCT02308878
Title: Executive Functioning in Heroin Users Following a Mobile Health Cognitive Stimulation Approach: a Randomized Controlled Trial
Brief Title: Mobile Health Cognitive Stimulation in Heroin Users
Acronym: Re@dict
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Gamito (Other)
Collaborators: Universidade Lusófona de Humanidades e Tecnologias (Other); Ares Do Pinhal-Associação De Recuperação De Toxicodependentes (Unknown)
Responsible Party: Sponsor-Investigator, Pedro Gamito, PhD (Full Professor), Universidade Lusófona de Humanidades e Tecnologias
Organization: Universidade Lusófona de Humanidades e Tecnologias (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLB_SUD01
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Substance Use Disorder
Keywords: Opioid Abuse Disorder; Cognitive Therapy; Executive Function; Mobile Health; Rehabilitation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment-as-usual (No Intervention): This group consists of treatment-as-usual for opioid dependence syndrome.
- Mobile health cognitive stimulation (Experimental): Cognitive stimulation using mobile technology with m-Health applications.
  Interventions: Behavioral: Mobile health cognitive stimulation

INTERVENTIONS:
Behavioral: Mobile health cognitive stimulation
  Arms: Mobile health cognitive stimulation

SUMMARY:
Heroin use has been related to brain dysfunction particularly in the prefrontal cortex. These effects are evident in neuropsychological impairments in attention, memory and executive functioning of heroin users. To assess these deficits and the application of a novel approach of cognitive stimulation to heroin users in treatment for opioid dependence, we have carried out a neuropsychological intervention program with mobile health technology. Patients diagnosed with opioid dependence were submitted to cognitive stimulation during four weeks in a three-day/week basis.

ELIGIBILITY:
Inclusion Criteria:

* Only patients that scored higher than the cutoff values for their age on the Mini Mental Examination Test and with no clinical scores on the Symptoms Checklist Revised will be included in the study.

Exclusion Criteria:

* Patients with alcohol dependence or with history of previous neurological disorders will be excluded from the study. Patients will be also screened for minimal computer literacy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-10; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in the results of Frontal Assessment Battery - FAB | 1 month
  The participants were assessed in frontal lobe functions at the beginning of the rehabilitation and after 10 rehabilitation sessions, which had the approximate duration of one month.

CONTACTS AND LOCATIONS:
Locations (1):
- Ares Do Pinhal-Associação De Recuperação De Toxicodependentes, Sintra, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided